CLINICAL TRIAL: NCT03511365
Title: Evaluation of Alterations in Serum Inflammatory Markers and Fecal Microbiota Following Administration of the Probiotic Formulation VSL#3 in Patients With Nonalcoholic Fatty Liver Disease
Brief Title: Effects of Probiotic on Inflammation and Microbiota in Patients With NASH
Acronym: NASHPro
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: IRB haulted the study there was no evidence that the probiotic would benefit the patient
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Bruce Hirsch, Assistant Professor of Medicine, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17-0514
Record Dates: First submitted 2018-04-06; First posted 2018-04-27 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Probiotics MeSH Descriptor Data 2018; Interleukin-17 MeSH Descriptor Data 2018
Keywords: Probiotic; Microbiome; Inflammation; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Inflammation

STUDY DESIGN:
Intervention Model Description: Single group interventional pilot study with each subject serving as his or her own control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic administration (Experimental): After baseline collection of serum and fecal microbiota, each subject will be administered the probiotic formulation VSL#3 450 Billion CFU Twice daily for 8 weeks. Serum and fecal microbiota will again be collected at the end of the intervention and compared with baseline with each subject serving as his or her own control.
  Interventions: Biological: Probiotic Formulation VSL#3

INTERVENTIONS:
Biological: Probiotic Formulation VSL#3 — Probiotic VSL#3 administration.

SUMMARY:
Individuals with clinically identified non-alcoholic fatty liver disease will undergo baseline evaluation of IL-17 and other inflammatory markers as well as microbiome determination. The probiotic formulation VSL#3 450 Billion CFU twice daily will be administered for 8 weeks and the determination of Il-17 and microbiome will be repeated. Each subject will serve as his or her own control.

DETAILED DESCRIPTION:
This study is designed as a prospective trial of the effects of probiotic on inflammatory and stool profiles in patients with NAFLD. These patients are actively followed by the Division of Hepatology. They will have confirmed normal liver function tests and absence of hepatitis C virus in order to be eligible for this study. Eligible subjects will be identified within the outpatient setting of the Division of Hepatology of the Northwell Health System.

Division of Hepatology 400 Community Drive Manhasset, NY 11030 516-562-4281

Candidate subjects will be identified by investigators as a part of their typical work flow. Subjects will be evaluated according to inclusion and exclusion criteria presented. Eligible patients will be provided with a packet containing study information and informed consent documents. Should a patient remain interested in study participation, informed consent will be obtained. Financial compensation will not be provided to subjects.

Forty patients with NAFLD will be enrolled.

Following enrollment and informed consent, subjects will undergo the following assessments:

1. Medical History Questionnaire
2. Current Medication List

Blood and stool samples will be obtained prior to study initiation and again after 8 weeks of exposure.

Protocol for biological sample collection:

Whole Blood Collection - Venipuncture will be performed under standard conditions. Three heparinized tubes will be obtained which each tube containing approximately 10 cc of whole blood Samples will be de-identified. Peripheral Blood Cells will be isolated from whole blood samples according to standard protocols.

Serum cytokine levels, including IL-10 and IL-17, will be assessed.

Stool Collection - Patients will be provided with stool collection kits. Samples will be de-identified. Stool samples will be preserved in a -20 degree freezer in the Division of Infectious Diseases.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Capable of giving informed consent
* Diagnosed with NAFLD as defined by the American Association for the Study of Liver Diseases (AASLD) who are treated or seen solely at the outpatient clinic at the Department of Hepatology at 400 Community Drive in Manhasset NY

Exclusion Criteria:

* Cirrhosis
* Absence of secondary causes of hepatic fat accumulation including:
* Excessive alcohol consumption
* Hepatitis C
* Wilson's Disease
* Lipodystrophy
* Starvation
* Parenteral Nutrition
* Abetalipoproteinemia
* Specific Medications: Amiodarone, Methotrexate, Tamoxifen, Corticosteroids, Valproate, Anti-retroviral agents)
* Reye's Syndrome
* HELLP Syndrome
* Inborn errors of metabolism (LCAT deficiency, cholesterol ester storage disease, Wolman disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Change in Il-17 levels with probiotic administration | 8 weeks
  Percent decrease in Il levels will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwell Health, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li J, Sung CY, Lee N, Ni Y, Pihlajamaki J, Panagiotou G, El-Nezami H. Probiotics modulated gut microbiota suppresses hepatocellular carcinoma growth in mice. Proc Natl Acad Sci U S A. 2016 Mar 1;113(9):E1306-15. doi: 10.1073/pnas.1518189113. Epub 2016 Feb 16. PMID 26884164